CLINICAL TRIAL: NCT01920464
Title: Place of Flixovate® in the Treatment Pathway and Its Conditions of Use in Infants Aged From 3 to 12 Months Between 2010 and 2012 by French GPs and Private Paediatricians
Acronym: flixovate HAS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116296
Record Dates: First submitted 2013-06-27; First posted 2013-08-12 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
this study has been request by french health authorities to evaluate the use of flixovate in infants and its place in the treatment pathway.

this study has 2 main pbjectives: 1/ Evaluation of changes in the prescription share of Flixovate® compared to other topical corticosteroids (low, medium and high potency) in the population of infants aged from 3 to 12 months, from 1st January 2010 to 31st December 2012. 2/Description of the conditions of use of Flixovate® in infants aged less than 12 months (infant profile, dosage form, dosage, treatment duration, prior, concomitant and subsequent treatments etc.).

ELIGIBILITY:
Inclusion Criteria:

Analysis of changes in share of prescriptions:

* Infants who received at least one prescription of topical steroids between 1st January 2010 and 31st December 2012.
* Infants aged 3 to 12 months on the day of prescription of topical steroids.

Description of the conditions of use and patient profiles:

* Infants who received at least one prescription of topical steroids between 1st January 2010 and 31st December 2012.
* Infants aged 3 to 12 months on the day of prescription of topical steroids.

Exclusion Criteria:

* none

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: retrospective database extraction
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Description of the conditions of use of Flixovate® in infants aged less than 12 months | baseline
  data collected and analysed: Profile of prescribers (age, sex, geographic location), Profile of infants (age, age group, gender, Z-score, medical history), Conditions (diagnoses corresponding to prescriptions of Flixovate®, dosage, mean duration of treatment and duration in classes, previous treatment, concomitant medications, treatments prescribed after discontinuation of Flixovate®. (emollients and other topical steroids).
- Evaluation of changes in the prescription share of Flixovate® compared to other topical corticosteroids (low, medium and high potency) in the population of infants aged from 3 to 12 months, from 1st January 2010 to 31st December 2012. | baseline, one year, 2 years, 3 years
  data collected and analysed: Profile of prescribers (age, gender, geographical location). Number of prescriptions of Flixovate® and other topical steroids by class, INN and brand name

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline